CLINICAL TRIAL: NCT00529503
Title: A Randomized Phase IIb Placebo-controlled Study of R-ICE Chemotherapy With and Without SGN-40 (Anti-CD40 Humanized Monoclonal Antibody) for Second-line Treatment of Patients With Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: A Randomized Phase IIb Placebo-Controlled Study of R-ICE Chemotherapy With and Without SGN-40 for Patients With DLBCL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SG040-0005
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin
Keywords: Lymphoproliferative Disorders; Lymphoma; Antigens, CD40; Antibody, Monoclonal; Combined Modality Therapy; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hematologic Diseases; Immunoproliferative Disorders; Lymphatic Diseases
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoproliferative Disorders; Lymphoma; Hematologic Diseases; Immunoproliferative Disorders; Lymphatic Diseases | interventions — dacetuzumab; Rituximab; Etoposide; Carboplatin; Ifosfamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): SGN-40, rituximab, etoposide, carboplatin, ifosfamide
  Interventions: Drug: SGN-40; Drug: rituximab; Drug: etoposide; Drug: carboplatin; Drug: ifosfamide
- 2 (Placebo Comparator): placebo, rituximab, etoposide, carboplatin, ifosfamide
  Interventions: Drug: placebo; Drug: rituximab; Drug: etoposide; Drug: carboplatin; Drug: ifosfamide

INTERVENTIONS:
Drug: SGN-40 — 2-8 mg/kg IV. Cycle 1: Days -1, 3, 8, 15; Cycles 2, 3: Days 1, 8, 15.
  Other Names: dacetuzumab
  Arms: 1
Drug: placebo — Volume as equivalent to corresponding SGN 40 dose IV. Cycle 1: Days -1, 3, 8, 15. Cycles 2, 3: Days 1, 8, 15.
  Arms: 2
Drug: rituximab — 375 mg/m2 IV. Cycle 1: Day -2; Cycles 2, 3: Day 1
  Other Names: Rituxan
Drug: etoposide — 100 mg/m2 IV. Cycles 1-3: Days 1, 2 and 3.
  Other Names: Toposar, Vepesid
Drug: carboplatin — AUC=5 mg/mL min IV. Cycles 1-3: Day 2.
  Other Names: Paraplatin
Drug: ifosfamide — 5 g/m2 24 hr. IV infusion. Cycles 1-3: Day2.
  Other Names: Ifex

SUMMARY:
This is a randomized trial to estimate the activity of R-ICE plus SGN-40 vs. R-ICE plus placebo in patients with DLBCL. The study will assess safety and tolerability and will measure any additional clinical benefit observed in patients receiving SGN-40.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of de novo or transformed DLBCL, or follicular grade 3b lymphoma.
* Received at least four cycles of first-line therapy with R-CHOP, or equivalent.
* Best clinical response to first-line therapy of stable disease, partial response, or complete response.
* At least one measureable lesion that is both greater than or equal to 1.5cm by radiographic imaging and by positive FDG-PET scan.

Exclusion Criteria:

* Leptomeningeal or central nervous system lymphoma.
* Received any therapy for relapsed or progressive disease except for local radiation, steroids, or rituximab.
* Received a hematopoietic stem cell transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Complete response as assessed by CT and PET scans and revised response criteria for malignant lymphoma. | 9 weeks

SECONDARY OUTCOMES:
Adverse events, laboratory values, and anti-drug antibody immune responses. | 9 weeks
Partial response, failure free survival, overall survival, and response for one and two years following treatment. | Every 3 months for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Drachman, MD, Study Director — Seagen Inc.
Locations (66):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Christiana Care Health Systems, Newark, Delaware
  - Georgetown University, Washington D.C., District of Columbia
  - MD Anderson Cancer Center, Orlando, Orlando, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Louisville - James Graham Brown Cancer Center, Louisville, Kentucky
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - San Juan Oncology Associates, Farmington, New Mexico
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor Sammons Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - MultiCare Health System, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia
- Australia (6):
  - St. Vincent's Hospital - Sydney, Darlinghurst, New South Wales
  - Gosford & Wyong Hospital, Gosford, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Royal Brisbane and Women's Hospital, Herston, Queensland
  - St. Vincent's Hospital, Melbourne, Fitzroy, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- Belgium (3):
  - Universite de Gent, Ghent
  - AZ Sint-Augustinus, Wilrijk
  - Cliniques Universitaires UCL de Mont-Goddine, Yvoir
- Czechia (3):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
- France (9):
  - Centre Hospitalier Andre Mignot, Le Chesnay
  - Centre Leon Berard - Centre regional de lutte contre le cancer Rhone-Alpes, Lyon
  - Hopital Hotel Dieu, Nantes
  - Groupe Hospitalier Necker - Enfants Malades, Paris
  - Hopitaux du Haut Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - Hematologie CHU Purpan, Toulouse
  - Institut Gustave-Roussy, Villejuif
- Germany (3):
  - Johannes-Gutenberg Universitat Mainz, Mainz
  - KH Maria Hilf-Franziskushaus, Mönchengladbach
  - Universitatsklinikum Ulm, Ulm
- Hungary (4):
  - Debreceni Egyetem Orvos - es Egeszsegtudomanyi Centrum, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, IInd Department of Internal Medicine, Győr
  - Kaposi Mor Oktato Korhaz, Kaposvár
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikat Kozpont, Szeged
- Italy (3):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Azienda Ospedaliera Universitaria Senese, Siena
- Poland (6):
  - Szpital Akademii Medycznej w Gdansku, Gdansk
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi, Lodz
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Centrum Onkologii Institut im. Marii Sklodowskiej-Curie, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1, Wroclaw
- Spain (5):
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Paul, Barcelona
  - H. Duran y Reynals Institue Catala D'Oncologia, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario La Fe, Valencia

REFERENCES:
- [Result] Fayad L, Ansell SM, Advani R, Coiffier B, Stuart R, Bartlett NL, Forero-Torres A, Kuliczkowski K, Belada D, Ng E, Drachman JG. Dacetuzumab plus rituximab, ifosfamide, carboplatin and etoposide as salvage therapy for patients with diffuse large B-cell lymphoma relapsing after rituximab, cyclophosphamide, doxorubicin, vincristine and prednisolone: a randomized, double-blind, placebo-controlled phase 2b trial. Leuk Lymphoma. 2015;56(9):2569-78. doi: 10.3109/10428194.2015.1007504. Epub 2015 Feb 26. PMID 25651427